CLINICAL TRIAL: NCT03009981
Title: A Phase 3 Study of Androgen Annihilation in High-Risk Biochemically Relapsed Prostate Cancer
Brief Title: A Study of Androgen Annihilation in High-Risk Biochemically Relapsed Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-19
Record Dates: First submitted 2017-01-03; First posted 2017-01-04 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: PSA; Degarelix; Apalutamide; Abiraterone Acetate; Radical Prostatectomy; Bicalutamide; Leuprolide; Lupron
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Gonadotropin-Releasing Hormone; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide; bicalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Degarelix Monotherapy OR Leuprolide/Bicalutamide (Active Comparator): Patients will receive degarelix OR leuprolide with bicalutamide.
  Interventions: Drug: LHRH Analogue
- Arm B: Degarelix/Apalutamide (Experimental): Patients will receive apalutamide and either degarelix OR leuprolide. Patients on this arm will NOT take bicalutamide at any point in the treatment course.
  Interventions: Drug: Apalutamide; Drug: LHRH Analogue
- Arm C: Degarelix/Apalutamide/Abiraterone/Prednisone (Experimental): Patients will receive apalutamide and abiraterone acetate, in addition to either degarelix OR leuprolide. Patients on this arm will NOT take bicalutamide at any point in the treatment course.
  Interventions: Drug: Apalutamide; Drug: LHRH Analogue; Drug: Abiraterone Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Apalutamide — Take apalutamide 240 mg (four 60 mg tablets) orally once daily, starting on C1D1 and continuing throughout 52-week treatment period.
  Other Names: Erleada
  Arms: Arm B: Degarelix/Apalutamide; Arm C: Degarelix/Apalutamide/Abiraterone/Prednisone
Drug: LHRH Analogue — Patients will receive a LHRH analogue therapy of either Degarelix OR Leuprolide with bicalutamide.
  Degarelix:
  Patients will receive subcutaneous injections every 28 days (+/- 3 days). Patients will receive a loading dose of 240 mg (two 120 mg injections) on C1D1, followed by maintenance dose of 80 mg on Day 1 of subsequent cycles.
  Leuprolide:
  Patients treated with leuprolide will receive a 7.5 mg IM injection on C1D1. Patients in arm A ONLY will take this in combination with bicalutamide 50 mg orally once daily starting on C1D1 and continuing for 28 days through completion of cycle 1. Starting on C2D1, patients will continue on one of the following two treatments at investigator discretion:
  1. Leuprolide 7.5 mg IM injection on Day 1 of subsequent cycles without concurrent bicalutamide.
     OR:
  2. Leuprolide 22.5 mg IM injection at the following visits without concurrent bicalutamide: C2D1, C5D1, C8D1, and C11D1.
  Other Names: Degarelix (Firmagon); Leuprolide (Lupron) and Bicalutamide
Drug: Abiraterone Acetate — Take abiraterone acetate 1000 mg (four 250 mg tablets) orally once daily, starting on C1D1 and continuing throughout 52-week treatment period.
  Other Names: Zytiga
  Arms: Arm C: Degarelix/Apalutamide/Abiraterone/Prednisone
Drug: Prednisone — Take two prednisone 5 mg tablets daily, starting on C1D1 and continuing throughout the 52-week treatment period. Following completion of treatment period, patients will taper off prednisone per institutional guidelines. Suggested tapering plan: prednisone 5 mg daily for 7 days, then 2.5 mg daily for 7 days before discontinuing.
  Other Names: Deltasone
  Arms: Arm C: Degarelix/Apalutamide/Abiraterone/Prednisone

SUMMARY:
This is a randomized, open-label, three-arm, phase 3 study in men with biochemically recurrent prostate cancer and PSA doubling time ≤ 9 months at the time of study entry.

DETAILED DESCRIPTION:
Patients will be stratified by PSA doubling time (< 3 months vs. 3-9 months) and randomized in 1:1:1 fashion to one of three treatment arms: (1) Control arm consisting of LHRH analogue monotherapy (degarelix or leuprolide), (2) Experimental arm consisting of apalutamide in combination with LHRH analogue, and (3) Experimental arm consisting of apalutamide, abiraterone acetate + prednisone, and LHRH analogue. Patients will be treated for a maximum duration of 52 weeks and then enter follow up phase until the time of PSA progression, development of metastasis, or patient withdrawal from study, whichever occurs first. Patients with PSA progression will be followed long term until the development of castration resistance, first metastasis, and death.

The primary endpoint of the study is PSA progression-free survival in the intent-to-treat patient population. PSA progression during the 52-week treatment period is defined as a rising PSA confirmed on repeat measurement, and at least 25% and 2 ng/mL above nadir or baseline, whichever is lower. PSA progression during follow up defined as PSA > 0.2 ng/mL confirmed by repeat measurement at least 2 weeks later. Secondary study endpoints include PSA progression-free survival in testosterone-evaluable population, 36-month PSA progression-free survival rate in both intent-to-treat and testosterone-evaluable populations, time to testosterone recovery, time to castration resistance, metastasis-free survival, quality of life, and safety. Each experimental arm will be compared against the control arm in pair-wise fashion. The study is not powered to detect differences in primary or secondary endpoints between the two experimental arms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* Prior radical prostatectomy
* Biochemically recurrent prostate cancer with PSA doubling time ≤ 9 months at the time of study entry. Calculation of PSA doubling time should include the use of all available PSA values obtained within past 6-12 months prior to randomization, with a minimum of 3 values separated by at least 2 weeks apart. PSA values obtained prior to therapeutic interventions (e.g. salvage radiation) will be excluded. PSA doubling time to be estimated using Memorial Sloan Kettering Cancer Center online calculator (https://www.mskcc.org/nomograms/prostate/psa-doubling-time)
* Prior adjuvant or salvage radiation or not a candidate for radiation based upon clinical assessment of disease characteristics and patient co-morbidities.
* Screening PSA > 0.5 ng/mL
* No definitive evidence of metastases on screening CT or MRI of abdomen/pelvis and radionuclide whole body bone scan per the judgment of the investigator. Abdominal and/or pelvic lymph nodes measuring 2 cm or less in short axis diameter are allowed. Lesions identified on other imaging modalities (e.g. PSMA or choline PET) that are not visualized on CT and/or MRI or radionuclide bone scan are allowed. Equivocal lesions on bone scan should be followed up with additional imaging as clinically indicated.
* Screening serum testosterone > 150 ng/dL
* Eastern Cooperative Oncology Group (ECOG) Performance Status grade 0 or 1
* Age ≥ 18 years
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to cycle 1 day 1
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Adequate organ function as defined by the following laboratory values at screening:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) < 2.5 x upper limit of normal (ULN)
  * Total serum bilirubin ≤1.5 x ULN. In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, subject may be eligible)
  * Serum potassium ≥ 3.5 mmol/L. Supplementation and re-screening is allowed.
  * Estimated creatinine clearance > 45 ml/min using Cockroft-Gault equation
  * Platelets ≥ 100,000/microliter independent of transfusion and/or growth factors within 3 months prior to randomization
  * Hemoglobin ≥ 9.0 g/dL independent of transfusion and/or growth factors within 3 months prior to randomization
  * Serum albumin ≥ 3.0 g/dL

Exclusion Criteria:

* Prior androgen deprivation therapy and/or first generation anti-androgen (e.g. bicalutamide, nilutamide, flutamide) for biochemically recurrent prostate cancer. Prior ADT and/or first generation anti-androgen in the (neo)adjuvant and/or salvage setting before, during, and/or following radiation or surgery is allowed provided last effective dose of ADT and/or first-generation anti-androgen is > 9 months prior to date of randomization and total duration of prior therapy is ≤ 36 months.
* Prior treatment with CYP17 inhibitor (e.g. ketoconazole, abiraterone acetate, galeterone) or second generation androgen receptor antagonist including apalutamide or enzalutamide
* Prior chemotherapy for prostate cancer except if administered in neoadjuvant or adjuvant setting
* Use of 5-alpha reductase inhibitor within 42 days prior to cycle 1 day 1
* Use of investigational agent within 28 days prior to randomization
* Use of other prohibited medications within 7 days prior to cycle 1 day 1 on study (Arms B and C only)
* Prior bilateral orchiectomy
* Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy)
* Uncontrolled hypertension
* Gastrointestinal disorder affecting absorption or the ability to swallow tablets
* Baseline severe hepatic impairment (Child-Pugh Class B & C)
* Intercurrent illness that is not controlled such as active infection, psychiatric illness/social situations that would limit compliance with study requirements
* Any chronic medical condition requiring a higher dose of corticosteroid than equivalent of 5 mg prednisone/prednisolone once daily

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
PSA progression-free survival in the intent-to-treat population | 36 months
  To compare PSA progression-free survival in each of the experimental arms (LHRH analogue + apalutamide; LHRH analogue + apalutamide +abiraterone acetate) versus the control arm (LHRH analogue) among all randomized patients (intent-to-treat population).

SECONDARY OUTCOMES:
PSA progression-free survival in the testosterone-evaluable population | 36 months
  Compare PSA progression-free survival in testosterone-evaluable population in each experimental arm versus the control arm. Testosterone-evaluable population includes all patients who achieve serum testosterone recovery to > 50 ng/dL with subsequent PSA measurements sufficient for evaluation
PSA progression-free survival in both the intent-to-treat and testosterone-evaluable populations | 36 months
  To compare the 36-month PSA progression-free survival rate in each experimental arm versus the control arm in both the intent-to-treat and testosterone-evaluable populations.
Serum testosterone | 12 months
  To compare the time to recovery of serum testosterone to greater than 50 ng/dL in each experimental arm versus the control arm.
Time to castration resistance | 6 years
  To compare the time to castration resistance in each experimental arm versus the control arm.
Metastasis-Free Survival | 6 years
  To compare metastasis-free survival in each experimental arm versus the control arm.
Overall Survival | 6 years
  To compare overall survival in each experimental arm versus the control arm.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 years
  To characterize the safety profile in each treatment arm
Quality of life Expanded Prostate Cancer Index Composite (EPIC) | 72 months
  Expanded Prostate Cancer Index Composite (EPIC)
Quality of life Hot Flash Daily Interference Scale (HFRDIS) | 72 months
  Hot Flash Daily Interference Scale (HFRDIS)
Quality of life EQ-5D-5L | 72 months
  EQ-5D-5L
Quality of life PROMIS Fatigue | 72 months
  PROMIS Fatigue
Quality-adjusted survival | 72 months
  To compare the quality-adjusted survival (overall survival multiplied by utility score) of patients in each experimental arm versus the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Evanthia Galanis, MD, Principal Investigator — Alliance Foundation Trials, LLC.; Rahul Aggarwal, MD, Study Chair — University of California, San Francisco
Locations (69):
- United States (69):
  - The Mayo Clinic - Phoenix, Phoenix, Arizona
  - Sharp Memorial Hospital, Chula Vista, California
  - City of Hope National Medical Center, Duarte, California
  - Palo Alto Medical Foundation, Fremont, California
  - VA Central California Health Care System, Fresno, California
  - Sharp Memorial Hospital, La Mesa, California
  - Palo Alto Medical Foundation, Mountain View, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - University of California San Diego - Moores Cancer Center, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Palo Alto Medical Foundation, Santa Cruz, California
  - Adventist Health St. Helena/St. Helena Hospital/Martin O'Neil Cancer Center, St. Helena, California
  - Palo Alto Medical Foundation, Sunnyvale, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Loyola University, Maywood, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Eastern Maine Medical Center, Brewer, Maine
  - New England Cancer Specialists, Kennebunk, Maine
  - New England Cancer Specialists, Scarborough, Maine
  - New England Cancer Specialists, Topsham, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute, Milford, Massachusetts
  - Dana Farber Cancer Institute, South Weymouth, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology & Hematology, Concord, New Hampshire
  - New Hampshire Oncology & Hematology, Hooksett, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, Middletown, New Jersey
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center- Cancer Center, Las Cruces, New Mexico
  - Christus St. Vincent's Regional Cancer Center, Santa Fe, New Mexico
  - VA Western New York, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Ctr - New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - VA Salisbury, Salisbury, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Dayton Physicians Miami Valley South, Centerville, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Toledo Clinic, Toledo, Ohio
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Spartanburg Medical Center/Gibbs Cancer Center, Spartanburg, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Marshfield Clinic Cancer Center, Marshfield, Wisconsin
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Zietman AL, Chung CS, Coen JJ, Shipley WU. 10-year outcome for men with localized prostate cancer treated with external radiation therapy: results of a cohort study. J Urol. 2004 Jan;171(1):210-4. doi: 10.1097/01.ju.0000100980.13364.a6. PMID 14665878
- [Background] Humphrey PA, Moch H, Cubilla AL, Ulbright TM, Reuter VE. The 2016 WHO Classification of Tumours of the Urinary System and Male Genital Organs-Part B: Prostate and Bladder Tumours. Eur Urol. 2016 Jul;70(1):106-119. doi: 10.1016/j.eururo.2016.02.028. Epub 2016 Mar 17. PMID 26996659
- [Background] Zelefsky MJ, Ben-Porat L, Scher HI, Chan HM, Fearn PA, Fuks ZY, Leibel SA, Venkatraman ES. Outcome predictors for the increasing PSA state after definitive external-beam radiotherapy for prostate cancer. J Clin Oncol. 2005 Feb 1;23(4):826-31. doi: 10.1200/JCO.2005.02.111. PMID 15681527
- [Background] Qu Y, Dai B, Ye D, Kong Y, Chang K, Jia Z, Yang X, Zhang H, Zhu Y, Shi G. Constitutively active AR-V7 plays an essential role in the development and progression of castration-resistant prostate cancer. Sci Rep. 2015 Jan 7;5:7654. doi: 10.1038/srep07654. PMID 25563505
- [Background] Gershon RC, Rothrock N, Hanrahan R, Bass M, Cella D. The use of PROMIS and assessment center to deliver patient-reported outcome measures in clinical research. J Appl Meas. 2010;11(3):304-14. PMID 20847477
- [Derived] Aggarwal R, Heller G, Hillman DW, Xiao H, Picus J, Taplin ME, Dorff T, Appleman L, Weckstein D, Patnaik A, Bryce A, Shevrin D, Mohler J, Anderson D, Rao A, Tagawa S, Tan A, Halabi S, Dooley K, O'Brien P, Chen R, Ryan CJ, Eggener SE, Morris MJ; EORTC-55994 Study Group. PRESTO: A Phase III, Open-Label Study of Intensification of Androgen Blockade in Patients With High-Risk Biochemically Relapsed Castration-Sensitive Prostate Cancer (AFT-19). J Clin Oncol. 2024 Apr 1;42(10):1114-1123. doi: 10.1200/JCO.23.01157. Epub 2024 Jan 23. PMID 38261983